CLINICAL TRIAL: NCT01292928
Title: Stenting of the Superficial Femoral (SFA) and Proximal Popliteal Arteries (PPA) With the Boston Scientific INNOVA Self-Expanding Bare Metal Stent System
Brief Title: SuperNOVA Clinical Stenting Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G100291
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Atherosclerosis of Native Arteries of the Extremities, Unspecified
Keywords: Atherosclerosis, Superficial Femoral Artery (SFA), Proximal Popliteal Artery (PPA), lower extremities, Stenting
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stent (Experimental): Stent implantation into SFA/PPA
  Interventions: Device: Stent implantation

INTERVENTIONS:
Device: Stent implantation — Stent implantation during the index procedure.

SUMMARY:
The primary objective of this clinical study is to determine whether the Innova Stent System shows acceptable performance in long-term (12-month) safety rates and vessel patency when treating femoropopliteal lesions.

DETAILED DESCRIPTION:
Atherosclerosis is a systemic disease that has become increasingly recognized in the expanding elderly population as a significant cause of morbidity and mortality. Atherosclerosis in the vessels of the lower extremities can cause a variety of symptoms ranging from intermittent claudication to ischemic rest pain and critical ischemia with major tissue loss. Typically, femoropopliteal lesions have been difficult to successfully treat with endovascular therapy because the disease is often diffuse and located in an area of the body subject to significant mobility stresses such as extension, contraction, compression, elongation, flexion and torsion.

The SuperNOVA clinical study is a prospective, single arm, controlled, multicenter, global study. Approximately 50 centers located in the United States, Europe, Canada and/or Australia are expected to participate in recruiting patients needing treatment of lesions in their femoropopliteal arteries. A maximum of 300 subjects will be enrolled to ensure that a minimum of 296 stented segments are treated with the Innova Stent System.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 and older
2. Chronic symptomatic lower limb ischemia defined as Rutherford categories 2, 3 or 4
3. Stenotic, restenotic (from angioplasty only) or occlusive lesion(s) located in the native superficial femoral artery or proximal popliteal artery:

   1. Degree of stenosis >/=70% by visual angiographic assessment
   2. Vessel diameter >/= 4 and </= 7mm
   3. Total lesion length (or series of lesions) >/=30mm and </= 190 mm (note: tandem lesions may be treated, provided that the tandem lesion segment can be covered with only one stent)
   4. If lesion is restenotic, PTA treatment must be >3 months prior to stent placement
   5. Target lesion located at least three centimeters above the inferior edge of the femur
4. Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (<50% stenosis) to the ankle or foot
5. Subject (or Legal Guardian) is willing and able to provide consent before any study-specific tests or procedures are performed and agrees to attend all required follow-up visits

Exclusion Criteria:

1. Previous stent placement in the target vessel
2. Subjects who have undergone prior surgery of the SFA/PPA in the target limb to treat atherosclerotic disease
3. Subjects who have undergone prior percutaneous transluminal angioplasty (PTA) in the target SFA/PPA in the past 3 months
4. Use of atherectomy devices or other adjunctive treatment in the SFA/PPA during the index procedure
5. History of major amputation in the same limb as the target lesion
6. Life expectancy less than 12 months due to other medical co-morbid condition(s) that could limit the subject's ability to participate in the clinical study, limit the subject's compliance with the follow-up requirements, or impact the scientific integrity of the clinical study
7. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated.
8. Intolerance to antiplatelet, anticoagulant, or thrombolytic medications
9. Platelet count <150,000 mm3 or >600,000 mm3
10. Concomitant renal failure with a serum creatinine >2.0 mg/dL
11. Receiving dialysis or immunosuppressant therapy
12. Pregnancy
13. Current participation in another investigational drug or device clinical study
14. Known allergy to Nitinol
15. Septicemia at the time of the index procedure
16. Presence of other hemodynamically significant outflow lesions requiring intervention within 30 days of the index procedure
17. Target lesion is within or near an aneurysm
18. Acute ischemia and/or acute thrombosis of the SFA/PPA
19. Persistent, intraluminal thrombus of the proposed target lesion post- thrombolytic therapy
20. Perforated vessel as evidenced by extravasation of contrast media
21. Heavily calcified lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Powell, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (49):
- United States (28):
  - Medical Center East, Birminham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Francis Medical Center, Peoria, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - Willis Knighton Bossier Medical Center, Bossier City, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Frederick Memorial Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Northern Michigan Hospital, Petoskey, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - St. Joseph's Hospital Health Center, Liverpool, New York
  - Mid-Carolina Cardiology Presbyterian Hospital, Charlotte, North Carolina
  - Rex Hospital, Raliegh, North Carolina
  - Coastal Surgery Specialists, Wilmington, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - UPMC - Passavant, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Methodist North Hospital, Memphis, Tennessee
  - St. Thomas Research Institute, LLC, Nashville, Tennessee
  - VA North Texas Health Care System, Dallas, Texas
  - Heart Center of Northe Texas, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Swedish Medical Center, Seattle, Washington
- Allgemeines Krankenhaus AKH, Vienna, Austria
- Belgium (5):
  - Imelda Ziekenhuis, Bonheiden
  - AZ Sint-Blasius, Campus Dendermonde, Dendermonde
  - Ziekenhuis Oost Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen
- Canada (4):
  - Fleurimont Hospital, Sherbrook, Quebec
  - Guelph General Hospital, Guelph
  - Hospital Maisonneuve-Rosemont, Montreal
  - Winnipeg Health Sciences Centre, Winnipeg
- Germany (4):
  - Center or Diagnostic Radiology and Minimally Invasive Therapy / Gefäßzentrum am JuedischenKrankenhaus, Berlin
  - Ev. Luth. Diakonissenanstalt Flensburg, Flensburg
  - Herzzentrum Leipzig GmbH/Park Krankenhaus, Leipzig
  - Friedrich-Ebert-Krankenhaus Neumuenster GmbH, Neumünster
- Japan (6):
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Tokeidai Memorial Hospital, Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki-shi, Hyōgo
  - Kishiwada Tokushukai Hospital, Kishiwada-shi, Osaka
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Morinomiya Hospital, Osaka
- Northern General Hospital, Sheffield, United Kingdom

REFERENCES:
- [Background] Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G; VIVA Physicians, Inc. Performance goals and endpoint assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. 2007 May 1;69(6):910-9. doi: 10.1002/ccd.21104. PMID 17377972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 299 subjects were enrolled and treated with the Innova™ Self-Expanding Stent System in this prospective, single-arm, non-randomized clinical study at 49 investigative centers in The Unites States, Canada, Japan and Europe, from 1 April 2011 to 28 June 2013 (with a temporary enrollment suspension from 13 May 2011 to 25 April 2012)
Groups:
- Innova Stent: Stent implantation into Superficial Femoral Artery (SFA) / Proximal Popliteal Artery (PPA)
Period: Overall Study
Arm/Group | Innova Stent
Started | 299
Completed 12-Month Clinical Follow-up | 266
Completed | 275
Not Completed | 24
Not completed — Death | 8
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- Innova Stent: Stent implantation into SFA/PPA
Arm/Group | Innova Stent
Number analyzed (Participants) | 299
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 222
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 4
  Caucasian | 238
  Asian (Japanese) | 42
  Black, or African heritage | 13
  Native Hawaiian or other Pacific Islander | 1
  American Indian or Alaska Native | 1
Region of Enrollment [Number; unit: participants]
  Canada | 31
  Austria | 6
  Belgium | 52
  United States | 117
  Japan | 42
  United Kingdom | 7
  Germany | 44
General Medical History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Smoking | 251
    Current Diabetes Mellitus | 121
    Medically-Treated Diabetes | 105
    History of Hyperlipidemia requiring medication | 224
    History of Hypertension requiring medication | 239
    History of Chronic Obstructive Pulmonary Disease | 25
Cardiac History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Coronary Artery Disease | 130
    History of Myocardial Infarction (MI) | 74
    History of Congestive Heart Failure | 25
    History of Percutaneous Coronary Intervention | 85
    History of Coronary Artery Bypass Graft Surgery | 54
    Stable Angina | 44
    Unstable Angina | 1
    No Angina | 245
Neurological/Renal History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Transient Ischemic Attacks | 21
    History of Cerebrovascular Accident | 24
    History of Renal Insufficiency | 31
    History of Renal Percutaneous Intervention | 4
Peripheral Vascular History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Peripheral Vascular Surgery | 27
    History of Other Peripheral Interventions | 125
    History of Claudication | 281
Baseline Lesion Characteristics: Treated Limb [Number; unit: lesions]
  Right leg | 138
  Left leg | 161
Baseline Lesion Characteristics: Reference Vessel Diameter [Mean (Standard Deviation); unit: millimeters] | 5.6 (0.7)
Baseline Lesion Characteristics: Diameter Stenosis [Mean (Standard Deviation); unit: percentage occluded] | 91.7 (9.2)
Baseline Lesion Characteristics: Target Lesion Length [Mean (Standard Deviation); unit: millimeters] | 90.8 (44.4)
Baseline Lesion Characteristics: Presence of Calcification [Number; unit: lesions]
  None/Mild | 88
  Moderate | 103
  Severe | 106
  Not Available | 2

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint and Components
Description: The safety endpoint assesses the occurrence of Major Adverse Events (MAEs) defined as all causes of death through 1 month, target limb major amputation through 12 months and/or target lesion revascularization through 12 months
Time Frame: 1 month for death, 12 months for target limb major amputation , and target lesion revascularization
Population: From the 275 subjects that were eligible for the 12-Month Follow-Up, data for the Primary Safety Endpoint were available for 268 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Innova Stent
Number analyzed (Participants) | 268
percentage of participants
  12-Month MAE-Free Rate | 85.8 [81.1 to 89.8]
  12-Month MAE (Composite Endpoint) | 14.2 [10.2 to 18.9]
  All Causes of Deaths at 1 Month | 0.0 [0.0 to 1.4]
  Target Limb Major Amputations | 0.4 [0.0 to 2.1]
  Target Lesion Revascularization | 14.2 [10.2 to 18.9]

2. Primary Outcome: Co-Primary Efficacy Endpoints
Description: The co-primary efficacy endpoints assess vessel primary patency at 12 months post-procedure.
  * The co-primary efficacy analysis (1) will assess vessel primary patency in stented segments intended to be treated with core matrix stents (20 to 150 mm).
  * The co-primary efficacy analysis (2) will assess vessel primary patency in stented segments intended to be treated with the entire stent matrix (20 to 200 mm).
Time Frame: 12 months
Population: From the 275 subjects that were eligible for the 12-Month Follow-Up, data for the Co-Primary Efficacy Endpoints were available for 268 subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Innova Stent Core Matrix (20-150 mm): Core Matrix Stent implantation into SFA/PPA
- Innova Stent Entire Matrix (20-200 mm): Entire Matrix Stent implantation into SFA/PPA
Arm/Group | Innova Stent Core Matrix (20-150 mm) | Innova Stent Entire Matrix (20-200 mm)
Number analyzed (Participants) | 231 | 268
percentage of participants | 69.7 [63.3 to 75.6] | 66.8 [60.8 to 72.4]

3. Secondary Outcome: Secondary Safety Endpoint and Components
Description: The secondary safety endpoint assesses the occurrence of Major Adverse Events (MAEs) through 30 days. MAEs will include all causes of death, target limb major amputation and/or target lesion revascularization through 1 month
Time Frame: 1 month
Population: From the 299 enrolled subjects, data for the Secondary Safety Endpoint was available for 297 subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Innova Stent
Number analyzed (Participants) | 297
percentage of participants
  1-Month MAE-Free Rate | 99.7 [98.1 to 100]
  1-Month MAE (Composite Endpoint) | 0.3 [0.0 to 1.9]
  All Causes of Deaths | 0.0 [0.0 to 1.2]
  Target Limb Major Amputation | 0.0 [0.0 to 1.2]
  Target Lesion Revascularization | 0.3 [0.0 to 1.9]

4. Other Pre Specified Outcome: Technical and Procedural Success
Description: * Technical success: ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30%
  * Procedural success: technical success with no MAEs within 24 hours of the procedure
Time Frame: Up to 24 hours after the procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Innova Stent
Number analyzed (Participants) | 299
percentage of participants
  Technical Success | 99 [97.1 to 99.8]
  Procedure Success | 99 [97.1 to 99.8]

5. Other Pre Specified Outcome: Primary Patency
Description: Primary patency is the percentage of lesions (target stented segments) that reach a time point without a hemodynamically significant stenosis assessed by Duplex Ultrasound (DUS) and without Target Lesion Revascularization (TLR) or bypass of the target lesion.
Time Frame: 12 months
Population: From the 275 subjects that were eligible for the 12-Month Follow-Up, data for the Primary Patency Analysis was available for 268 subjects/lesions
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Innova Stent
Number analyzed (Participants) | 268
Number analyzed (Lesions) | 268
percentage of lesions | 66.8 [60.8 to 72.4]

6. Other Pre Specified Outcome: Assisted Primary Patency
Description: Assisted primary patency is the percentage of lesions without TLR and those with TLR (not due to complete occlusion or bypass) that reach a time point without restenosis.
Time Frame: 12 months
Population: From the 275 subjects that were eligible for the 12-Month Follow-Up, data for the Assisted Primary Patency Analysis was available for 256 subjects
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Innova Stent
Number analyzed (Participants) | 256
percentage of lesions | 83.6 [78.5 to 87.9]

7. Other Pre Specified Outcome: Stent Fracture Rate
Description: Vascular InterVentional Advances (VIVA) definitions:
  Grade 0: No strut fractures
  Grade I: single strut fracture
  Grade II: multiple strut fractures
  Grade III: stent fracture(s) with preserved alignment of the components
  Grade IV: stent fracture(s) with mal-alignment of the components
  Grade V: stent fracture(s) in a trans-axial spiral configuration
Time Frame: 12 months
Population: From the 276 subjects that were eligible for the 12-Month Follow-Up, data for the Stent Fracture Analysis were available for 250 subjects
Measure: Number; unit: percentage of stents
Units Other Than Participants: stents
Arm/Group | Innova Stent
Number analyzed (Participants) | 250
Number analyzed (stents) | 264
percentage of stents
  Grade II | 0.76
  Grade III | 1.14
  Grade IV | 0.38
  Total | 2.27

8. Other Pre Specified Outcome: Rutherford Classification
Description: Class 0: Asymptomatic
  Class 1: Mild claudication
  Class 2: Moderate claudication
  Class 3: Severe claudication
  Class 4: Ischemic rest pain
  Class 5: Minor tissue loss - nonhealing ulcer, focal gangrene with diffuse pedal edema
  Class 6: Major tissue loss - extending above metatarsal (MT) level
  Rate of Primary Sustained Clinical Improvement: an improvement in Rutherford classification of one or more categories as compared to pre-procedure without the need for repeat TLR.
  Rate of Secondary Sustained Clinical Improvement: an improvement in Rutherford classification of one or more categories as compared to pre-procedure including those subjects with repeat TLR.
  Rate of Clinical Deterioration: downgrade in Rutherford classification of one or more categories as compared to pre-procedure
Time Frame: 12 months
Population: From the 275 subjects that were eligible for the 12-Month Follow-Up, data for the Rutherford Classification Analysis was available for 263 subjects
Measure: Number; unit: percentage of participants
Arm/Group | Innova Stent
Number analyzed (Participants) | 263
percentage of participants
  Rutherford Class 0 | 65.8
  Rutherford Class 1 | 19.0
  Rutherford Class 2 | 8.0
  Rutherford Class 3 | 6.8
  Rutherford Class 4 | 0.0
  Rutherford Class 5 | 0.4
  Rutherford Class 6 | 0.0
  Primary Sustained Clinical Improvement | 79.5
  Secondary Sustained Clinical Improvement | 90.1
  Clinical Deterioration | 2.7
  No Change from Baseline | 7.2

9. Other Pre Specified Outcome: Rate of Hemodynamic Improvement
Description: The Ankle-Brachial Index (ABI) is the ratio between the systolic pressure measured at the ankle and the systolic pressure measured in the arm.
  Hemodynamic Improvement: Increases in ABI of ≥ 0.10 or to an ABI ≥ 0.90 as compared to pre-procedure without the need for repeat TLR.
  Hemodynamic Improvement (Including TLR): Increases in ABI of ≥0.10 or to an ABI ≥0.90 as compared to pre-procedure including TLR.
Time Frame: 12 months
Population: 278 subjects were included in the Rate of Hemodynamic Improvement Analysis (275 subjects eligible for the 12-Month Follow-Up + 3 subjects with TLR)
Measure: Number; unit: percentage of limbs
Units Other Than Participants: limbs
Arm/Group | Innova Stent
Number analyzed (Participants) | 278
Number analyzed (limbs) | 278
percentage of limbs
  Hemodynamic Improvement | 59
  Hemodynamic Improvement (Including TLR) | 68.3

10. Other Pre Specified Outcome: Walking Improvement Assessed by the Walking Impairment Questionnaire
Description: The Walking Impairment Questionnaire (WIQ) is a validated functional assessment questionnaire that evaluates walking ability with regard to speed, distance and stair climbing ability as well as the reasons that walking ability might be limited. Range of scores is between 0% and 100% with 100% being the best and 0% being the worst score.
Time Frame: 12 months
Population: From the 275 subjects that were eligible for the 12-Month Follow-Up, data for the Walking Improvement assessed by the Walking Impairment Questionnaire were available for 265 subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innova Stent
Number analyzed (Participants) | 265
units on a scale
  Walking Impairment | 73.87 (30.98)
  Change from Baseline | 34.03 (37.22)

11. Other Pre Specified Outcome: Walking Improvement (Time) Assessed by 6 Minute Hall Walk
Description: Assessment of walking improvement (time) by the administration of the 6 Minute Walk Test (6MWT). Participants were asked to walk for as long as they could; up to 6 minutes.
Time Frame: 12 months
Population: From the 275 subjects that were eligible for the 12-Month Follow-Up, data for the Walking Improvement Assessed by 6 minute Hall Walk Analysis were available for 246 subjects
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Innova Stent
Number analyzed (Participants) | 246
minutes
  Baseline | 5.5 (1.3)
  12-Months | 5.7 (0.9)

12. Other Pre Specified Outcome: Walking Improvement (Distance) Assessed by 6 Minute Hall Walk
Description: Assessment of walking improvement (distance) by the administration of the 6 Minute Walk Test (6MWT). Participants were asked to walk for as long as they could; up to 6 minutes.
Time Frame: 12 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Innova Stent
Number analyzed (Participants) | 246
meters
  Baseline | 278.6 (119.1)
  12-Months | 358.9 (147.2)

13. Other Pre Specified Outcome: Quality of Life
Description: Improved Quality of Life assessed by the SF-36 Health Survey. The validated SF-36 Survey, where scores are calibrated so that 50 is the average score or norm, was utilized (scores ranging from 0, worst possible health to 100, best possible health). The SF-36 is a multipurpose, proprietary health survey with 36 questions that yield eight health component scales that can be further summarized into two summary scores: mental and physical health scores. The eight health component scales that can be computed from the questionnaire are physical function, role-physical, bodily pain, general health, vitality, role-emotional, mental health and social functioning.
Time Frame: 12 months
Population: From the 275 subjects that were eligible for the 12-Month Follow-Up, data for the Quality of Life Analysis were available for 265 subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innova Stent
Number analyzed (Participants) | 265
units on a scale
  Physical Functioning | 41.17 (11.38)
  Physical Functioning Change from Baseline | 6.53 (10.29)
  Role Physical | 43.39 (11.48)
  Role Physical Change from Baseline | 5.14 (11.9)
  Role Emotional | 45.45 (13.22)
  Role Emotional Change from Baseline | 3.49 (14.61)
  Social Functioning | 48.12 (10.55)
  Social Functioning Change from Baseline | 2.66 (13.26)
  Bodily Pain | 46.52 (11.33)
  Bodily Pain Change from Baseline | 7.28 (12.19)
  Mental Health | 50.19 (10.46)
  Mental Health Change from Baseline | 2.33 (11.21)
  Vitality | 50.57 (10.98)
  Vitality Change from Baseline | 3.10 (10.68)
  General Health Perceptions | 44.65 (9.9)
  General Health Perceptions Change from Baseline | 1.32 (9.51)
  Mental Component Score | 51.14 (10.71)
  Mental Component Score Change from Baseline | 0.86 (11.69)
  Physical Component Score | 42.66 (10.30)
  Physical Component Score Change from Baseline | 6.31 (10.23)

ADVERSE EVENTS:
Time Frame: 12 months
Description: From the 276 subjects that were eligible for the 12-Month Follow-Up, data for the Adverse Events Analysis were available for 266 subjects
Arm/Group | Innova Stent
Serious Adverse Events (participants affected / at risk) | 143/266
Other Adverse Events (participants affected / at risk) | 116/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Innova Stent (N=266)
Acute coronary syndrome (Cardiac disorders) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 3 (3)
Angina pectoris (Cardiac disorders) | 6 (7)
Angina unstable (Cardiac disorders) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (4)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Administration site conditions: Catheter site haemorrhage (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Administration site conditions: Impaired healing (General disorders) | 2 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (1)
Allergic oedema (Immune system disorders) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Enterocolitis bacterial (Infections and infestations) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4)
Postoperative wound infection (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 (4)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 1 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Marasmus (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (3)
Convulsion (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 4 (6)
Arterial thrombosis limb (Vascular disorders) | 5 (6)
Circulatory collapse (Vascular disorders) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 47 (59)
Femoral artery occlusion (Vascular disorders) | 11 (17)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
liac artery stenosis (Vascular disorders) | 7 (8)
Intermittent claudication (Vascular disorders) | 18 (24)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (4)
Peripheral embolism (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Vulval abscess (Infections and infestations) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Innova Stent (N=266)
Intermittent claudication (Vascular disorders) | 24 (27)
Catheter site haematoma (General disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Femoral artery stenosis (Vascular disorders) | 18 (20)
Haematoma (Vascular disorders) | 6 (7)
Vascular procedure complication (Injury, poisoning and procedural complications) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish the Results, provided that before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any Confidential Information or other proprietary information of Sponsor from the proposed publication or presentation.